CLINICAL TRIAL: NCT00480220
Title: Specific Care and Assistance Plan for Alzheimer's Disease: Impact Study on Disease Progression and Management Modalities
Brief Title: Specific Care and Assistance Plan for Alzheimer's Disease
Acronym: PLASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0200601; PHRC (Other Grant/Funding Number: 2001 and 2006)
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
Keywords: specific care; assistance plan; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Specific Intervention as Global care and support program
  Interventions: Procedure: Global care and support program
- 2 (No Intervention): 'No specific intervention'

INTERVENTIONS:
Procedure: Global care and support program
  Arms: 1

SUMMARY:
The main objective of this work is to assess the feasibility and efficacy of a specific Care and Assistance Plan for Alzheimer's disease (PLASA). The main outcome measure selected is incapacity in carrying out the basic activities of daily living, evaluated by the ADCS-ADL scale .

The PLASA was developed by a working group appointed by the Direction Générale de la Santé as part of the government programme of action on Alzheimer's disease (October 2001, Ministère de l'Emploi et de la Solidarité).

DETAILED DESCRIPTION:
It is estimated that at the present time about 50% of dependence in the elderly is related to dementias. Alzheimer's disease is the most common of these, and there are 100 000 new cases in France every year (Girard Report). Very often, once the diagnosis has been established these persons do not receive regular, codified follow-up, whereas Alzheimer's disease is a chronic disease which progresses over several years and leads to a variety of complications which must be identified and managed.

The main objective of this work is to assess the feasibility and efficacy of a specific Care and Assistance Plan for Alzheimer's disease (PLASA). The main outcome measure selected is incapacity in carrying out the basic activities of daily living, evaluated by the ADCS-ADL scale .

The PLASA was developed by a working group appointed by the Direction Générale de la Santé as part of the government programme of action on Alzheimer's disease (October 2001, Ministère de l'Emploi et de la Solidarité).

Methods The multicentre prospective study will be randomised within each centre. Study population: 1200 patients will be recruited in 20 French university hospitals and 40 general hospitals.

Inclusion criteria: Patients presenting mild to moderate Alzheimer's disease diagnosed by the NINCDS-ADRDA criteria (MMSE between 12 and 26), living at home and with an identified principal caregiver.

Randomisation and patient follow-up: After randomisation within each centre (specialised department of the university or general hospital), half of the patients will be managed according to the PLASA (group A). The other patients will receive the usual management of the centres (group B).

The PLASA includes detailed evaluation of the patient's cognitive and non-cognitive function, regular and standardised follow-up, management of complications and the setting up of assistance and support services according to common guidelines. As part of the PLASA, patients will be systematically seen in consultation every six months.

Data collection: In group A, data will be collected during six-monthly consultations for the duration of the study (T0, T6, T12, T18, T24). In group B, data will be collected during consultations at T0, T12 and T24. The coordinating centre (Toulouse) will contact every 6 months (T6, T12, T18, T24), by post or by telephone, the principal caregiver for collection of intermediate data in both groups. These data include evaluation of activities of daily living (ADCS-ADL), utilization of support and care services (RUD ), as well as subjective assessment of disease severity (ADCS-CGIC ). The patient's quality of life will also be evaluated in both groups at T0, T12 and T24.

Statistical analysis: 1200 subjects are needed to reveal a 30% decrease in incapacities in activities of daily living in the group of patients followed according to the PLASA.

Bivariate analysis will be carried out using the standard tests for this type of study (chi-squared test and Student's t test). The efficacy of the PLASA will be assessed by multivariate analysis, taking potential confounders into account.

Expected results: This project should contribute to better long-term management of patients with Alzheimer's disease and should reduce the burden on families.

ELIGIBILITY:
Inclusion Criteria:

* patient seen in consultation in one of the centres participating in the study
* patient with probable or possible AD according to NINCDS-ADRDA criteria
* patient with an MMSE score between 12 and 26 (mild to moderate disease)
* patient capable of understanding and responding to the evaluations made
* patient who is not confined to bed or chair
* patient living at home with an informal caregiver
* informed consent of the patient (or legal representative) and of the caregiver agreeing to take part in the study.

Exclusion Criteria:

* patient with an MMSE score of less than 12 or over 26
* patient incapable of understanding and responding to the evaluations made
* patient confined to bed or chair
* patient living at home without an informal carer or in an institution
* patient with a concomitant disorder threatening the vital prognosis at two years
* patient with a dementia other than AD
* patient already included in another research programme.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2003-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of the specific care and assistance plan for Alzheimer's disease in a study randomised within each centre. The main aim of the care plan is to reduce loss of independence. | 2 years

SECONDARY OUTCOMES:
Impact of the care and assistance plan: - on the mode of the patient's admission to an institution - on utilization of assistance, support and healthcare services (RUD questionnaire) - and on overall clinical evaluation of change (ADCS-CGIC). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: VELLAS Bruno, PD PhD, Study Director — University Hospital, Toulouse
Locations (40):
- France (40):
  - Hospital, Albi
  - Hospital Center, Alès
  - University Hospital, Angers
  - Hospital, Annecy
  - Hospital Center, Bar-le-Duc
  - University Hospital, Brest
  - Hospital Center, Carcassonne
  - Service de Gérontologie, Carvin
  - Hospital, Chambéry
  - Georges Clémenceau Hospital, Champcueil
  - Hospital Center, Grasse
  - University Hospital, Grenoble
  - Hôpital Charles Foix - La Triade, Ivry-sur-Seine
  - Hospital Center, Lannemezan
  - Hospital Center, Lavaur
  - Hospital, Lens
  - University Hospital, Lille
  - Hospital Center, Louviers
  - University Hospital, Lyon
  - University Hospital Sainte Marguerite, Marseille
  - University Hospital, Montpellier
  - University Hospital, Nice
  - Hospital Center, Niort
  - University Hospital, Nîmes
  - Hospital Bichat - Claude Bernard, Paris
  - Hospital Center Notre Dame du Bon Secours, Paris
  - University Hospital BROCA - La Rochefoucauld, Paris
  - University Hospital Pitié-Salpétrière, Paris
  - University Hospital Sainte Perrine, Paris
  - Hospital center, Plaisir
  - University Hospital, Reims
  - Hospital Center, Roubaix
  - University Hospital, Rouen
  - Hospital Center, Saint-Dizier
  - Hospital Center, Sézanne
  - University Hospital, Hôpital Xavier Arnozan, Toulouse
  - University Hospital, Toulouse
  - Hospital, Valenciennes
  - Hospital Center, Villejuif
  - Hospital, Wasquehal

REFERENCES:
- [Background] Callahan CM, Boustani MA, Unverzagt FW, Austrom MG, Damush TM, Perkins AJ, Fultz BA, Hui SL, Counsell SR, Hendrie HC. Effectiveness of collaborative care for older adults with Alzheimer disease in primary care: a randomized controlled trial. JAMA. 2006 May 10;295(18):2148-57. doi: 10.1001/jama.295.18.2148. PMID 16684985
- [Background] Teri L, Gibbons LE, McCurry SM, Logsdon RG, Buchner DM, Barlow WE, Kukull WA, LaCroix AZ, McCormick W, Larson EB. Exercise plus behavioral management in patients with Alzheimer disease: a randomized controlled trial. JAMA. 2003 Oct 15;290(15):2015-22. doi: 10.1001/jama.290.15.2015. PMID 14559955
- [Background] Teri L, Logsdon RG, McCurry SM. Nonpharmacologic treatment of behavioral disturbance in dementia. Med Clin North Am. 2002 May;86(3):641-56, viii. doi: 10.1016/s0025-7125(02)00006-8. PMID 12168563
- [Background] Vickrey BG, Mittman BS, Connor KI, Pearson ML, Della Penna RD, Ganiats TG, Demonte RW Jr, Chodosh J, Cui X, Vassar S, Duan N, Lee M. The effect of a disease management intervention on quality and outcomes of dementia care: a randomized, controlled trial. Ann Intern Med. 2006 Nov 21;145(10):713-26. doi: 10.7326/0003-4819-145-10-200611210-00004. PMID 17116916
- [Derived] Nourhashemi F, Andrieu S, Gillette-Guyonnet S, Giraudeau B, Cantet C, Coley N, Vellas B; PLASA Group. Effectiveness of a specific care plan in patients with Alzheimer's disease: cluster randomised trial (PLASA study). BMJ. 2010 Jun 3;340:c2466. doi: 10.1136/bmj.c2466. PMID 20522656
- [Derived] Nourhashemi F, Gillette-Guyonnet S, Andrieu S, Rolland Y, Ousset PJ, Vellas B; PLASA group. A randomized trial of the impact of a specific care plan in 1120 Alzheimer's patients (PLASA Study) over a two-year period: design and baseline data. J Nutr Health Aging. 2008 Apr;12(4):263-71. doi: 10.1007/BF02982632. PMID 18373036